CLINICAL TRIAL: NCT00929136
Title: The Effect of Regional Inflammation on Metabolism and Insulin Sensitivity in the Lower Extremity.
Brief Title: Peripheral Effects of Endotoxin on Insulin Resistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Niels Moller M.D. and Mads Buhl, M.D, University of Aarhus
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: Aarhus University Hospital
Record Dates: First submitted 2009-06-22; First posted 2009-06-26 (Estimated); Last update posted 2010-10-04 (Estimated); Status verified 2010-10

CONDITIONS: Healthy
Keywords: Endotoxin; Insulin resistance; Lipolysis; Proteolysis; Intracellular Insulin Signaling; Regional effects of inflammation/endotoxin
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endotoxin (Experimental)
  Interventions: Biological: USP endotoxin

INTERVENTIONS:
Biological: USP endotoxin — Continuous intra-arterial infusion
  Other Names: USP Endotoxin, LOT: G3E069

SUMMARY:
The aim of the study is to isolate the direct effects of endotoxin on glucose, lipid and protein metabolism. Eight healthy volunteers are enrolled. The hypothesis is that endotoxin will induce insulin resistance, lypolysis and proteolysis acutely.

ELIGIBILITY:
Inclusion Criteria:

1. Normal health
2. 22 < BMI < 28
3. Written Informed Concent

Exclusion Criteria:

1. Any disease
2. Any use of medication
3. Recent immobilization of a lower extremity

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
glucose concentration | 360 minutes observation

SECONDARY OUTCOMES:
Regional arteriovenous amino-acid balance | measured at t=180 and 360 minutes
Intra-cellular insulin signaling | measured at t=0, 120, and, 210 minutes
Regional arteriovenous lipid balance | measured at t=180 and 360 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Mads Buhl, M.D., Principal Investigator — Medical Department M (Endocrinology and Diabetes), Århus University Hospital, Denmark; Niels Moller, M.D., professor, Dmsc, Study Director — Medical Department M (Endocrinology and Diabetes), Aarhus University Hospital, Denmark
Locations (1):
- The Medical Research Laboratories, Dept. M, Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Buhl M, Bosnjak E, Vendelbo MH, Gjedsted J, Nielsen RR, K-Hafstrom T, Vestergaard ET, Jessen N, Tonnesen E, Moller AB, Pedersen SB, Pilegaard H, Bienso RS, Jorgensen JO, Moller N. Direct effects of locally administered lipopolysaccharide on glucose, lipid, and protein metabolism in the placebo-controlled, bilaterally infused human leg. J Clin Endocrinol Metab. 2013 May;98(5):2090-9. doi: 10.1210/jc.2012-3836. Epub 2013 Mar 29. PMID 23543661